CLINICAL TRIAL: NCT03659760
Title: Does Light and Noise Isolation Change the Melatonin Levels and Inflammatory Response After Cranial Surgery in an Intensive Care Unit
Brief Title: : Association of Melatonin Levels and Light and Noise Isolation in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Arik, Specialist in Anesthesia, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EmineMelatonin
Record Dates: First submitted 2018-08-31; First posted 2018-09-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cranial Nerve Diseases
Keywords: Melatonin; Interleukin; Transcranial; Surgery; Intensive care
MeSH Terms: conditions — Cranial Nerve Diseases

STUDY DESIGN:
Intervention Model Description: prospective randomize
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Isolated (Experimental): Group Isolated (Group II) (eyes closed with patch and ear plugged; between 24:00-06:00)
  Interventions: Other: Group Isolated
- Group Disrupted (No Intervention): Group Disrupted (Group I) (exposed to ambient light and noise)

INTERVENTIONS:
Other: Group Isolated — Eyes closed with patch and ears plugged between 24:00-06:00
  Arms: Group Isolated

SUMMARY:
Melatonin is secreted from the epiphyseal gland with a circadian rhythm and is known to be anti-inflammatory.

In this study, it is planned to investigate the effect of sleep disruptions on melatonin levels and inflammation parameters in intensive care patients underwent transcranial surgery

DETAILED DESCRIPTION:
Patients with Glasgow coma scale (GKS) >14, American Society of Anesthesiologist (ASA) I-III, intensive care patients underwent transcranial surgery will be included

Patients will be randomly allocated by a computer generated random numbers list into two groups.

Patients with sleep disruptions (Group I) (exposed to ambient light and noise) and Patients without sleep disruptions (Group II) (eyes closed with patch and ear plugged; between 24:00-06:00)

Melatonin levels will be measured by urine 6-sulfatoxymelatonin (a-MT6) levels, which is a product of melatonin degradation at 07:00 am preoperative and postoperative day 1 and day 3.

Plasma Interleukin-1 (IL-1), Interleukin- 6 (IL-6),C-reactive protein (CRP) levels will be measured at 07:00 am preoperative and postoperative day 1and day 3.

ELIGIBILITY:
Inclusion Criteria

* ASA 1-3
* Glasgow Coma Scale(GCS) >14

Exclusion Criteria:

* Glasgow Coma Scale(GCS) <14
* Patients who do not understand the questions, not awake
* Patient who treated with hormones
* Patient with infection or inflammatory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Melatonin level | At preoperative 07:00 am
  Melatonin will be measured urine 6-sulphatoxymelatonin
Melatonin level | 07:00 am postoprative day 1
  Melatonin will be measured urine 6-sulphatoxymelatonin
Melatonin level | 07:00 am postoprative day 3
  Melatonin will be measured urine 6-sulphatoxymelatonin

SECONDARY OUTCOMES:
IL-1,IL-6,CRP | : at 7 o'clock in the morning preoperative day, 7 in the morning on the first postoperative day and 7 in the morning on the third postoperative day hour
  serum

CONTACTS AND LOCATIONS:
Overall Officials: Emine Arık, Principal Investigator — Dr
Locations (1):
- Universty of Health Sciences, Dıskapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grima NA, Rajaratnam SMW, Mansfield D, Sletten TL, Spitz G, Ponsford JL. Efficacy of melatonin for sleep disturbance following traumatic brain injury: a randomised controlled trial. BMC Med. 2018 Jan 19;16(1):8. doi: 10.1186/s12916-017-0995-1. PMID 29347988
- [Background] Yasar NF, Badak B, Canik A, Bas SS, Uslu S, Oner S, Ates E. Effects of Sleep Quality on Melatonin Levels and Inflammatory Response after Major Abdominal Surgery in an Intensive Care Unit. Molecules. 2017 Sep 12;22(9):1537. doi: 10.3390/molecules22091537. PMID 28895895
- [Background] Osier N, McGreevy E, Pham L, Puccio A, Ren D, Conley YP, Alexander S, Dixon CE. Melatonin as a Therapy for Traumatic Brain Injury: A Review of Published Evidence. Int J Mol Sci. 2018 May 22;19(5):1539. doi: 10.3390/ijms19051539. PMID 29786658
- [Background] Kurdi MS, Patel T. The role of melatonin in anaesthesia and critical care. Indian J Anaesth. 2013 Mar;57(2):137-44. doi: 10.4103/0019-5049.111837. PMID 23825812